CLINICAL TRIAL: NCT02530905
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Titration, Safety, Tolerability, and Pharmacokinetics Study Followed by an Open-Label Safety and Efficacy Evaluation of SRP-4045 in Advanced-Stage Patients With Duchenne Muscular Dystrophy Amenable to Exon 45 Skipping
Brief Title: Dose-Titration and Open-label Extension Study of SRP-4045 in Advanced Stage Duchenne Muscular Dystrophy (DMD) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4045-101
Record Dates: First submitted 2015-08-10; First posted 2015-08-21 (Estimated); Results first posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-04

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Exon Skipping
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — casimersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (double-blind dose titration) (Placebo Comparator): Participants with genotypically confirmed Duchenne muscular dystrophy (DMD) characterized by deletions amenable to exon 45 skipping will receive placebo-matching to casimersen intravenous (IV) infusions, once weekly over approximately 12 weeks in the double-blind period.
  Interventions: Drug: Placebo
- SRP-4045 (double-blind dose titration) (Experimental): Participants with genotypically confirmed DMD characterized by deletions amenable to exon 45 skipping will receive weekly IV infusions of casimersen at four escalating dose levels, each for at least 2 weeks: 4 milligrams per kilograms (mg/kg) during Week 1 to Week 2, followed by 10 mg/kg during Week 3 to Week 4, followed by 20 mg/kg during Week 5 to Week 6, followed by 30 mg/kg beginning at Week 7 and continue over approximately Week 12 in the double-blind period.
  Interventions: Drug: SRP-4045
- SRP-4045 (open label extension period) (Experimental): All participants who completed double blind period will be enrolled to receive casimersen 30 mg/kg once weekly, for up to Week 144 in the open label extension period.
  Interventions: Drug: SRP-4045

INTERVENTIONS:
Drug: SRP-4045 — SRP-4045 solution for IV infusion.
  Arms: SRP-4045 (double-blind dose titration); SRP-4045 (open label extension period)
Drug: Placebo — SRP-4045 placebo-matching solution for IV infusion.
  Arms: Placebo (double-blind dose titration)

SUMMARY:
This is a first-in-human dose-titration and open-label extension study to assess safety, tolerability, and pharmacokinetics of SRP-4045 in advanced-stage Duchenne muscular dystrophy (DMD) patients with deletions amenable to exon 45 skipping.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled dose-titration study to assess safety, tolerability, and pharmacokinetics of 4 dose levels of SRP-4045 in genotypically confirmed advanced-stage DMD patients with deletions amenable to exon 45 skipping.

After completion of the dose-titration portion of the study and SRP-4045 is determined to be safe, all patients will be evaluated on open-label SRP-4045 for the duration of the study.

Safety, including adverse event monitoring, routine laboratory assessments, and cardiac testing will be monitored through the duration of the dose-titration and open-label portions of the study.

Clinical efficacy will be assessed at regularly scheduled study visits via quality of life questionnaires and tests of pulmonary and upper extremity function through the duration of the dose-titration and open-label portions of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Genotypically confirmed DMD (amenable to exon 45 skipping).
* Stable cardiac and pulmonary function.
* Limited or no ambulation.
* On a stable dose of oral corticosteroids for at least 24 weeks OR has not received corticosteroids for at least 24 weeks.

Exclusion Criteria:

* Current or previous treatment with the experimental agents SMT C1100 (BMN-195) or PRO045.
* Other experimental treatment in the past 12 weeks.
* If on cardiac medication, must be on a stable dose for the past 12 weeks.
* Major surgery within the past 3 months.

Other inclusion/exclusion criteria apply.

Ages: 7 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (3):
- United States (3):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 sites in United States.
Pre-assignment Details: Study conducted in 2 parts: Part 1 (Double-Blind Period [DBP]) and Part 2 (Open Label Extension Period [OLEP]). When Part 1 was completed and cumulative safety data was reviewed by an independent Data Safety Monitoring Board (DSMB), Part 2 was conducted.
Groups:
- Double-Blind Period: Placebo: Participants with genotypically confirmed Duchenne muscular dystrophy (DMD) characterized by deletions amenable to exon 45 skipping received placebo-matched to casimersen intravenous (IV) infusions, once weekly over approximately 12 weeks in the double-blind period.
- Double-Blind Period: Casimersen: Participants with genotypically confirmed DMD characterized by deletions amenable to exon 45 skipping received weekly IV infusions of casimersen at four escalating dose levels, each for at least 2 weeks: 4 milligrams per kilograms (mg/kg) during Week 1 to Week 2, followed by 10 mg/kg during Week 3 to Week 4, followed by 20 mg/kg during Week 5 to Week 6, followed by 30 mg/kg beginning at Week 7 and continued over approximately Week 12 in the double-blind period.
- Open Label Extension Period: Casimersen: All participants who completed double blind period were enrolled to receive casimersen 30 mg/kg once weekly, for up to Week 144 in the open label extension period.
Period: Double-Blind Period (12 Weeks)
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Casimersen | Open Label Extension Period: Casimersen
Started | 4 | 8 | 0
Received 4 mg/kg | 0 | 8 | 0
Received 10 mg/kg | 0 | 8 | 0
Received 20 mg/kg | 0 | 8 | 0
Received 30 mg/kg | 0 | 8 | 0
Completed | 4 | 8 | 0
Not Completed | 0 | 0 | 0
Period: Open Label Extension Period (132 Weeks)
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Casimersen | Open Label Extension Period: Casimersen
Started | 0 | 0 | 12 (All participants from the double-blind period amenable to exon 45 skipping were enrolled to open-label extension period.)
Completed | 0 | 0 | 11
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all randomized participants who received at least 1 dose of study drug (casimersen or placebo) in double-blind period.
Groups:
- Double-Blind Period: Placebo: Participants with genotypically confirmed DMD characterized by deletions amenable to exon 45 skipping received placebo-matched to casimersen IV infusions, once weekly over approximately 12 weeks in the double-blind period.
- Double-Blind Period: Casimersen: Participants with genotypically confirmed DMD characterized by deletions amenable to exon 45 skipping received weekly IV infusions of casimersen at four escalating dose levels, each for at least 2 weeks: 4 mg/kg during Week 1 to Week 2, followed by 10 mg/kg during Week 3 to Week 4, followed by 20 mg/kg during Week 5 to Week 6, followed by 30 mg/kg beginning at Week 7 and continued over approximately Week 12 in the double-blind period.
- Total: Total of all reporting groups
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Casimersen | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.0 (2.16) | 14.4 (3.29) | 13.6 (3.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 7 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse event (AE) was any untoward medical occurrence in a clinical trial participant, which does not necessarily have a causal relationship with the investigational drug. AEs also included abnormal physical examination findings (Physical examination were conducted per protocol and any clinically significant abnormal findings were recorded in medical history if pre-existing or addressed as an AE if new or worsening). TEAEs was defined as AEs that started, worsened, or became serious on or after the start of first infusion through 148 weeks. Number of participants with TEAEs were reported.
Time Frame: Baseline up to Week 148
Population: Safety set included all randomized participants who received at least 1 dose of study drug (casimersen or placebo) in both double-blind and open-label extension periods.
Measure: Count of Participants; unit: Participants
Groups:
- Double-Blind Period: Casimersen 4 mg/kg: Participants with genotypically confirmed DMD characterized by deletions amenable to exon 45 skipping received casimersen IV infusions, at a dose level of 4 mg/kg once weekly for 2 weeks (i.e. Week 1 to Week 2) in the double-blind period.
- Double-Blind Period: Casimersen 10 mg/kg: Participants with genotypically confirmed DMD characterized by deletions amenable to exon 45 skipping received casimersen IV infusions, at a dose level of 10 mg/kg once weekly for 2 weeks (i.e. Week 3 to Week 4) in the double-blind period.
- Double-Blind Period: Casimersen 20 mg/kg: Participants with genotypically confirmed DMD characterized by deletions amenable to exon 45 skipping received casimersen IV infusions, at a dose level of 20 mg/kg once weekly for 2 weeks (i.e. Week 5 to Week 6) in the double-blind period.
- Double-Blind Period: Casimersen 30 mg/kg: Participants with genotypically confirmed DMD characterized by deletions amenable to exon 45 skipping received casimersen IV infusions, at a dose level of 30 mg/kg once weekly from Week 7 to Week 12 in the double-blind period.
- Open Label Extension Period: Casimersen 30 mg/kg: All participants who completed double blind period were enrolled to receive casimersen 30 mg/kg once weekly, for up to Week 144 in the open label extension period.
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8 | 12
Participants | 4 | 5 | 3 | 3 | 7 | 12

2. Primary Outcome: Number of Participants With Potentially Clinically Significant (PCS) Laboratory Abnormalities Reported as TEAEs
Description: Laboratory parameters included serum chemistry (hepatic chemistry and renal chemistry), hematology, coagulation, and urinalysis. Number of participants with potentially clinically significant abnormal finding were reported as TEAEs. The Investigator determined whether abnormal assessment results were potentially clinically significant or not. Potentially clinical significance was defined as any variation in assessment results that had medical relevance resulting in an alteration in medical care.
Time Frame: Baseline up to Week 148
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8 | 12
Participants
  Serum chemistry: Hepatic chemistry | 0 | 0 | 0 | 0 | 0 | 0
  Serum chemistry: Renal chemistry | 0 | 0 | 0 | 0 | 0 | 0
  Hematolgy: Leukocytes | 0 | 0 | 0 | 0 | 2 | 4
  Hematolgy: Neutrophils | 0 | 0 | 0 | 0 | 4 | 6
  Coagulation: Platelet count | 0 | 0 | 0 | 0 | 2 | 2
  Urinalysis | 0 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities in Vital Signs Reported as TEAEs
Description: Vital sign parameters included systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), and body temperature. Number of participants with at least one potentially clinically significant abnormal vital signs findings were reported as TEAEs. The Investigator determined whether abnormal assessment results were potentially clinically significant or not. Potential clinical significance was defined as any variation in assessment results that had medical relevance resulting in an alteration in medical care.
Time Frame: Baseline up to Week 148
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8 | 12
Participants | 0 | 0 | 0 | 0 | 1 | 1

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities in Electrocardiogram (ECG) Reported as TEAEs
Description: Twelve-lead ECGs were performed at a consistent time of day throughout the study. Electrocardiograms were performed only after the participant was in the supine position, resting, and quiet for a minimum of 15 minutes. The ECG was manually reviewed and interpreted by medically qualified personnel. Number of participants with potentially clinically significant abnormalities in ECG reported as TEAEs were presented here. The Investigator determined whether abnormal assessment results were potentially clinically significant or not.
Time Frame: Baseline up to Week 148
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 1

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities in Echocardiograms (ECHO)
Description: Standard, 2-dimensional ECHOs were performed at a consistent time of day throughout the study.The ECHO was reviewed and interpreted by medically qualified personnel. Number of participants with potentially clinically significant abnormalities in ECHO were reported.
Time Frame: Baseline up to Week 148
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Casimersen
Description: Maximum Concentration (Cmax) of casimersen in plasma was evaluated.
Time Frame: Pre-infusion, 5 to 10 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16, and 24 hours post-dose at Weeks 1 (for 4 mg/kg ), 3 (for 10 mg/kg arm), 5 (for 20 mg/kg arm), 7 (for 30 mg/kg arm) in DBP and Week 60 (for 30 mg/kg arm) in OLEP
Population: Pharmacokinetic (PK) set included all randomized participants who received the planned full dose of study drug (casimersen) and for whom there are adequate PK samples from which to estimate PK parameters. Data was not planned to be collected and analyzed for placebo arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 12
Nanogram per milliliter (ng/mL) | 13700 (25.0) | 39400 (11.7) | 64400 (27.4) | 119000 (33.6) | 115000 (31.5)

7. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Casimersen
Description: Time to reach maximum plasma concentration (Tmax) of casimersen was evaluated.
Time Frame: as for outcome 6
Population: PK set included all randomized participants who received the planned full dose of study drug (casimersen or placebo) and for whom there are adequate PK samples from which to estimate PK parameters. Data was not planned to be collected and analyzed for placebo arm.
Measure: Median (Full Range); unit: Hour
Arm/Group | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 12
Hour | 1.11 [0.92 to 1.22] | 1.03 [0.93 to 1.17] | 1.03 [0.83 to 1.22] | 0.94 [0.83 to 1.18] | 0.95 [0.78 to 1.08]

8. Secondary Outcome: Area Under Concentration-time Curve From Time of Dosing to the Last Measurable Concentration (AUClast) of Casimersen in Plasma
Description: Area under the concentration-time curve from time zero to the last quantifiable concentration of casimersen in plasma were evaluated.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 12
Hour*nanogram per milliliter (hr*ng/mL) | 23100 (29.5) | 59500 (16.2) | 101000 (17.7) | 188000 (27.4) | 182000 (33.8)

9. Secondary Outcome: Area Under Concentration-Time Curve From Time Zero Pre-dose to Twenty-Four Hours Post-dose (AUC0-24) of Casimersen in Plasma
Description: Area under concentration-time curve from time zero pre-dose to twenty-four hours post-dos of casimersen in plasma were evaluated.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 12
h*ng/mL | 23200 (29.4) | 59500 (16.1) | 101000 (17.7) | 188000 (27.4) | 182000 (33.8)

10. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero Extrapolated to the Infinity (AUCinf) of Casimersen in Plasma
Description: Area under the concentration-time curve from time zero extrapolated to the infinity of casimersen in plasma was evaluated.
Time Frame: as for outcome 6
Population: PK set included all randomized participants who received the planned full dose of study drug (casimersen or placebo) and for whom there are adequate PK samples from which to estimate PK parameters. Here, "Overall number of participants analyzed" = number of participants evaluable for this outcome. Data was not planned to be collected and analyzed for placebo arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 12
h*ng/mL | 23300 (29.5) | 58300 (16.0) | 101000 (17.7) | 189000 (27.5) | 182000 (33.9)

11. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss) of Casimersen
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution at steady state of casimersen was evaluated.
Time Frame: as for outcome 6
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per kilogram (L/kg)
Arm/Group | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 12
Liter per kilogram (L/kg) | 0.369 (24.4) | 0.343 (12.5) | 0.407 (23.4) | 0.319 (31.4) | 0.367 (28.9)

12. Secondary Outcome: Elimination Half-life (T1/2) of Casimersen
Description: T1/2 is the time measured for the plasma concentration of drug to decrease by one half. T1/2 of casimersen was evaluated.
Time Frame: as for outcome 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 12
Hour | 2.92 (0.985) | 3.29 (0.640) | 3.71 (0.616) | 3.82 (0.741) | 3.45 (0.359)

13. Secondary Outcome: Total Clearance (CL) of Casimersen
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. CL of casimersen was evaluated.
Time Frame: as for outcome 6
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour per kilogram (L/h/kg)
Arm/Group | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 12
Liters per hour per kilogram (L/h/kg) | 0.177 (29.1) | 0.181 (15.9) | 0.205 (18.5) | 0.163 (27.7) | 0.180 (35.0)

14. Secondary Outcome: Mean Residence Time Extrapolated to Infinity (MRTinf) of Casimersen
Description: MRTinf = AUMCinf/AUCinf - T/2, where T was the infusion duration, and AUMCinf was the area under the first moment curve from time 0 extrapolated to infinite time, calculated using the linear/log trapezoidal method. MRTinf of casimersen was evaluated.
Time Frame: as for outcome 6
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 12
Hour | 2.08 (13.5) | 1.89 (16.1) | 1.98 (12.7) | 1.96 (16.6) | 2.04 (10.3)

15. Secondary Outcome: Double-Blind Period: Renal Clearance (CLR) of Casimersen
Description: Renal clearance was calculated using the partial AUC0-24 from the non-compartmental analysis in plasma and AE0-24. AUC0-24 was defined as area under the plasma concentration-time curve, from time 0 to 24 hours after completion of dosing. AE0-24 was defined as total cumulative amount excreted from 0 to 24 hours. Summarized data of all urine collection intervals are reported.
Time Frame: 0 to 4, 4 to 8, 8 to 12, and 12 to 24 hours post-dose at Weeks 1 (for 4 mg/kg ), 3 (for 10 mg/kg arm), 5 (for 20 mg/kg arm), 7 and 12 (for 30 mg/kg arm) in double-blind period
Population: PK set included all randomized participants who received the planned full dose of study drug (casimersen or placebo) and for whom there are adequate PK samples from which to estimate PK parameters. Here, "Overall number of participants analyzed"= number of participants evaluable for this outcome. Data was not planned to be collected and analyzed for placebo and open-label extension period arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/kg
Arm/Group | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg
Number analyzed (Participants) | 8 | 8 | 7 | 8
L/h/kg | 0.137 (25.8) | 0.162 (22.6) | 0.209 (29.0) | 0.177 (34.2)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Week 148
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Casimersen 4 mg/kg | Double-Blind Period: Casimersen 10 mg/kg | Double-Blind Period: Casimersen 20 mg/kg | Double-Blind Period: Casimersen 30 mg/kg | Open Label Extension Period: Casimersen 30 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8 | 0/8 | 0/8 | 1/8 | 3/12
Other Adverse Events (participants affected / at risk) | 4/4 | 5/8 | 3/8 | 3/8 | 7/8 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Period: Placebo (N=4) | Double-Blind Period: Casimersen 4 mg/kg (N=8) | Double-Blind Period: Casimersen 10 mg/kg (N=8) | Double-Blind Period: Casimersen 20 mg/kg (N=8) | Double-Blind Period: Casimersen 30 mg/kg (N=8) | Open Label Extension Period: Casimersen 30 mg/kg (N=12)
Septic embolus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Period: Placebo (N=4) | Double-Blind Period: Casimersen 4 mg/kg (N=8) | Double-Blind Period: Casimersen 10 mg/kg (N=8) | Double-Blind Period: Casimersen 20 mg/kg (N=8) | Double-Blind Period: Casimersen 30 mg/kg (N=8) | Open Label Extension Period: Casimersen 30 mg/kg (N=12)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 4
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 9
Tinea versicolour (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 3 | 4
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Urine calcium (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Drug withdrawal headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Device dislocation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 2
Thrombosis in device (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 3
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Application site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Application site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Application site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Catheter site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Delayed puberty (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The most restrictive relevant agreement provides that the PI can only publish the study results with the approval of Sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT02530905/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT02530905/SAP_001.pdf